CLINICAL TRIAL: NCT07358910
Title: Risk Assessment of Community Spread of Multiple Endemic Infectious Diseases in a One Health Perspective
Acronym: RACSMEI
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur du Cambodge (Other)
Collaborators: Institut Pasteur (Industry); CDC - Ministry of Health of Cambodia (Unknown); UMR ASTRE (CIRAD) (Unknown); Malaria Consortium (Other); Ministry of Agriculture, Forestry and Fisheries Cambodia (Unknown)
Responsible Party: Sponsor
Other Study IDs: IPasteurCambodge; 312353/Z/24/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Dengue; Chikungunya; Zika Virus Infection; Japanese Encephalitis; West Nile Virus; Tick-borne Encephalitis (TBE); Severe Fever With Thrombocytopenia Syndrome; Nipah Virus Infection; Hantavirus Infections; Hepatitis E; Brucellosis; Q Fever; Leptospirosis; Melioidosis; Influenza A and B; Malaria; Yellow Fever; Mayaro Fever; Usutu Virus Infection; Oropouche Fever; Rift Valley Fever; Arenavirus Infections; Measles; Mumps; Rubella; Human Papilloma Virus (HPV); Rotavirus Disease; Pertussis; Diphteria; Tetanus; Varicella; Hepatitis A; Norovirus Infections; Enterovirus; Adenovirus; Rhinovirus; Parvovirus; Respiratory Syncytial Virus (RSV); Cytomegalovirus; Epstein Barr Virus; Salmonella Typhi; Vibrio Cholerae; Legionella Pneumophila Pneumonia; Mycoplasma; Chlamydia; Lymphatic Filariasis; Toxoplasma Gondii; Giardiasis; Entamoeba Histolytica; Leishmaniasis; Strongyloides Stercoralis Infection; Ascaris Lumbricoides; Trichuris Trichiura; Clonorchis Sinensis; Opisthorchis Viverrini; Schistosomiasis; Streptococcus Pneumoniae; Meningitis
Keywords: Infectious disease; One Health; Population-based survey; Nationally representative survey; Seroepidemiology; Multiplex serology; Seroprevalence; Vector-borne diseases; Zoonoses; Vaccine-preventable diseases; Neglected tropical diseases; Transmission dynamics; Force of infection; Mathematical modelling; Spatial epidemiology; Precision public health; Cambodia
MeSH Terms: conditions — Dengue; Chikungunya Fever; Zika Virus Infection; Encephalitis, Japanese; Encephalitis, Tick-Borne; Severe Fever with Thrombocytopenia Syndrome; Henipavirus Infections; Hantavirus Infections; Hepatitis E; Brucellosis; Q Fever; Leptospirosis; Melioidosis; Malaria; Yellow Fever; Bunyaviridae Infections; Rift Valley Fever; Arenaviridae Infections; Measles; Mumps; Rubella; Rotavirus Infections; Whooping Cough; Tetanus; Chickenpox; Hepatitis A; Caliciviridae Infections; Enterovirus Infections; Adenoviridae Infections; Parvoviridae Infections; Epstein-Barr Virus Infections; Mycoplasma Infections; Chlamydia Infections; Elephantiasis, Filarial; Giardiasis; Leishmaniasis; Trichuriasis; Schistosomiasis; Meningitis; Communicable Diseases; Vector Borne Diseases; Zoonoses; Vaccine-Preventable Diseases; Neglected Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Human serum aliquots derived from venous blood collected in dry tubes and stored at ≤-80 °C for multiplex serology. In selected workflows, pathogen nucleic acids may be generated for testing but are not retained.
  Co-located animal specimens include sera (poultry, pigs, dogs, cattle, sheep/goats) and oral/rectal swabs; rodent specimens collected near households for laboratory testing. These samples are processed and archived according to standardized procedures. Environmental specimens retained include surface swabs, water samples (with 0.2 µm filtrates/membranes), air and soil samples from high-risk human-animal-environment interfaces. Vector collections (mosquito specimens obtained with BG-traps) are retained for entomological and pathogen investigations. All retained specimens are aliquoted as appropriate and stored in the IPC biobank under controlled temperatures for up to 15 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Human Community Cohort (National Population Sample): Probability-based, multi-stage population sample of ~10,000 participants (2-75 years old) recruited across urban and rural communities nationwide. Data include standardized questionnaires (demography, health conditions, mobility, animal contact, healthcare access) and serum biospecimens for multiplex serology;

SUMMARY:
RACSMEI addresses the high burden of infectious diseases in low- and middle-income countries, including Cambodia, where limited surveillance and laboratory capacity often obscure etiologies and transmission dynamics. This knowledge gap hinders the design of effective prevention and control strategies.

RACSMEI will improve understanding across multiple pathogens using a multidisciplinary One Health approach. We will answer key questions on burden, ecology, transmission and population immune status to inform targeted and culturally appropriate interventions. The project combines a nationally representative One Health survey, social-science methods, and multiplex, diverse diagnostics to efficiently test for 57 priority pathogens, including zoonotic and vector-borne agents, vaccine-preventable and elimination-targeted diseases, enteric, respiratory, and environmentally transmitted pathogens and selected neglected tropical diseases and parasites relevant to Cambodia.

Mathematical modelling will reconstruct and forecast transmission dynamics and assess the potential impact of future public-health strategies. By integrating intersectoral data and innovative methods, RACSMEI will generate actionable evidence for public-health authorities, support precision One Health interventions, and help reduce disease burden in affected communities. The project also aims to ensure the transferability of methods and insights to other countries facing similar challenges.

DETAILED DESCRIPTION:
RACSMEI is a nationwide, One Health, multi-pathogen initiative designed to generate integrated evidence for public-health decision-making in Cambodia. Beyond producing epidemiological findings, the project will establish a structured biobank and curated datasets intended to support long-term collaborative research, knowledge sharing, and evidence-informed policy. The program includes capacity building and technology transfer to strengthen national institutions and foster regional scientific leadership and international collaboration. Engagement with communities and national stakeholders is planned to facilitate future studies and promote the uptake of results in practice. Overall, RACSMEI aims to provide a scalable model for integrated infectious-disease assessment in low- and middle-income settings, creating durable infrastructure, partnerships, and decision-support resources that can be used beyond the project period.

ELIGIBILITY:
Inclusion Criteria:

* Residency in the village for more than 6 months;
* Age between 2 and 75 years old at the time of inclusion;
* For adults: provision of written consent;
* For children aged 2-17 years: written parental consent form, verbal assent from children aged 13-17 years;

Exclusion Criteria:

* Unable to understand or consent;
* Under guardianship or deprived of liberty;
* Medical conditions that impede survey participation;
* Refusal to participate in the study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises approximately 10,000 participants aged 2 to 75 years, drawn from 4,160 households across Cambodia's 25 provinces. Households will be randomly selected from 104 villages to ensure a nationally representative sample that reflects the country's diverse geographic and demographic characteristics. Participants will provide detailed socio-demographic information, enabling post-stratification weighted analysis of the sample's structure by sex, age, and geographic area to facilitate the extrapolation of findings to the entire population, ensuring that the study's conclusions are broadly applicable.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-04-16 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence of antibodies against an established panel of priority pathogens in the surveyed human populations: | At the time of blood sampling during household visits, over the inclusion period from December 2025 to April 2026.
  The proportion of sampled individuals with detectable antibodies against this priority panel of pathogens, measured using multiplex serological assays.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Flamand, Ph.D., Principal Investigator — Institut Pasteur du Cambodge
Locations (1):
- Institut Pasteur du Cambodge, Phnom Penh, Phnom Penh, Cambodia

REFERENCES:
- See also: Dedicated website page related to the study — https://www.pasteur-kh.org/racsmei/
- See also: Wellcome Trust project description page — https://wellcome.org/research-funding/funding-portfolio/funded-grants/racsmei-risk-assessment-community-spread-multiple